CLINICAL TRIAL: NCT04554875
Title: Derivation and Validation of a Scoring System to Distinguish Cryptococcosis and Adenocarcinoma in Pulmonary Nodules: a Multicenter Observational Study.
Brief Title: Derivation and Validation of a Scoring System to Distinguish Cryptococcosis and Adenocarcinoma in Pulmonary Nodules
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: 20200410
Record Dates: First submitted 2020-08-11; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Cryptococcosis; Lung Adenocarcinoma
MeSH Terms: conditions — Cryptococcosis; Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: Derivation Cohort of a Scoring System to Distinguish Cryptococcosis and Adenocarcinoma in Pulmonary Nodules
- Cohort 2: One of Validation Cohorts of a Scoring System to Distinguish Cryptococcosis and Adenocarcinoma in Pulmonary Nodules
  Interventions: Diagnostic Test: A scoring system
- Cohort 3: One of Validation Cohorts of a Scoring System to Distinguish Cryptococcosis and Adenocarcinoma in Pulmonary Nodules
  Interventions: Diagnostic Test: A scoring system
- Cohort 4: One of Validation Cohorts of a Scoring System to Distinguish Cryptococcosis and Adenocarcinoma in Pulmonary Nodules
  Interventions: Diagnostic Test: A scoring system

INTERVENTIONS:
Diagnostic Test: A scoring system — The scoring system was used to rate score patients.
  Groups: Cohort 2; Cohort 3; Cohort 4

SUMMARY:
Pulmonary cryptococcosis often manifests as isolated or multiple nodules, easily mimicking lung cancer clinically and radiologically, which ascribes the poor sensitivity of Cryptococcus culture and rarely positive of Cryptococcal antigen test in the absence of disseminated disease. Therefore, the aim of this study was to develop a predictive scoring system from the perspective of available clinical indicators, to differentiate cryptococcosis from adenocarcinoma in pulmonary nodules, which might be beneficial for the delicacy management of pulmonary nodules.

DETAILED DESCRIPTION:
Nodule is generally defined as a small, approximately spherical in morphology, circumscribed focus of abnormal tissue on computed tomography (CT) and no greater than 3cm in maximum diameter. Pulmonary nodules are not uncommon. A systematic review of CT screening lung cancer trials noted that a lung nodule was detected in up to 51% of study participants. More than 95% of detected nodules are benign and have a wide variety of causes, including infections, granulomatous disease, hamartomas, arteriovenous malformations, round atelectasis, and lymph nodes.

Pulmonary cryptococcosis is caused by Cryptococcus spp., a ubiquitous budding yeast-like basidiomycete that is endemic in many countries. Previously, Pulmonary cryptococcosis was thought to be an important opportunistic invasive mycosis in immunocompromised patients, such as AIDS, immunosuppressor used after organ transplantation, but it is also common in immunocompetent patients. Pulmonary cryptococcosis often manifests as isolated or multiple nodules, easily mimicking lung cancer clinically and radiologically, which ascribes the poor sensitivity of Cryptococcus culture and rarely positive of Cryptococcal antigen test in the absence of disseminated disease.

Therefore, the aim of this multicenter observational study was to develop a predictive scoring system from the perspective of available clinical indicators, to differentiate cryptococcosis from adenocarcinoma in pulmonary nodules, which might be beneficial for the delicacy management of pulmonary nodules.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulmonary nodules
* Evidence of pathological diagnosis for cryptococcosis or adenocarcinoma
* Data on high-resolution computed tomography (HRCT)

Exclusion Criteria:

* Pulmonary nodules greater than 3cm in maximum diameter
* Lack of data on HRCT

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pulmonary nodules, no greater than 3cm in maximum diameter, finally diagnosed with cryptococcosis or adenocarcinoma were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Area under receiver operating characteristic curve | up to 24 weeks
  Area under Receiver Operating Characteristic (ROC) curve was used to identify the diagnostic value of the scoring system.

SECONDARY OUTCOMES:
Sensitivity of the scoring system | up to 24 weeks
  Sensitivity of the scoring system was used to assess the true positive rate of pulmonary cryptococcosis
Specificity of the scoring system | up to 24 weeks
  Specificity of the scoring system was used to assess the true negative rate of pulmonary cryptococcosis

CONTACTS AND LOCATIONS:
Overall Officials: Jin-fu Xu, MD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai pulmonary hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided